CLINICAL TRIAL: NCT06340204
Title: Weekly Irinotecan Liposomes in Recurrent or Refractory Ewing Sarcoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University Shougang Hospital (Other); Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Tang Xiaodong, M.D., Head of Musculoskeletal Tumor Center, Peking University People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-EWS-03
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Ewing Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric (Experimental): pediatric patients
  Interventions: Drug: Irinotecan Hydrochloride Liposome Injection
- Adults (Experimental): Adult patients
  Interventions: Drug: Irinotecan Hydrochloride Liposome Injection

INTERVENTIONS:
Drug: Irinotecan Hydrochloride Liposome Injection — Irinotecan Hydrochloride Liposome Injection is given weekly by 5 doses every 6 weeks (5/6 qw).
  Other Names: duo en yi

SUMMARY:
The investigators explored the safety and activity of weekly irinotecan liposomes in patients with relapsed and metastatic Ewing Sarcoma.

DETAILED DESCRIPTION:
After standard multimodal therapy, the prognosis of relapsed and metastatic Ewing Sarcoma is dismal and unchanged over the last decades. The anti-tumor activity of irinotecan was demonstrated by several studies in the past. However, longer schedule of irinotecan infusion (traditionally dx5x2) has impacted quality of life in these patients. The irinotecan liposomes may be more active than the parent compound irinotecan since its ability to stay longer in circulation system, and much more convenient to given weekly.

Thus, the investigators explored the safety and activity of weekly irinotecan liposomes in patients with relapsed and metastatic Ewing Sarcoma after the failure of first-line chemotherapy with doxorubicin, vincristine, cyclophosphamide, ifosphamide and etoposide. Bayesian Optimal Interval (BOIN) design is adopted in this dose-finding study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Ewing sarcoma
* Evidence of Ewing sarcoma translocation by fluorescence in situ hybridization (FISH) or real-time polymerase chain reaction (RT-PCT).
* Recurrent or refractory tumors with no known curative treatment options according to the judgment of the investigator.
* Prior treatment consisted of standard Ewing Sarcoma chemotherapy agents including doxorubicin, vincristine, cyclophosphamide, ifosfamide and etoposide; metastatic relapsed and unresectable progressive disease (PD).
* Life expectancy of ≥ 3 months.
* Eastern Cooperative Oncology Group performance status 0-1.
* Measurable disease on CT or MRI by RECIST 1.1.
* Adequate organ function.
* Time elapsed from previous therapy must be ≥ 3 weeks for systemic therapy, ≥ 2 weeks for radiation therapy or major surgery.
* Patients who have undergone autologous hematopoietic stem cell transplantation are eligible once they have recovered from all toxicities from therapy.
* Patients who have received allogeneic hematopoietic stem cell transplantation will be eligible 6 months after the procedure provided there is no evidence of active graft-versus-host disease and immunosuppressive treatment has been discontinued for at least 30 days.
* Patients with central nervous system disease are eligible for enrollment if they have received prior radiotherapy or surgery to sites of central nervous system metastatic disease, have been off glucocorticoids for at least 4 weeks, have no overt evidence of neurological deficit and are ≥ 6 weeks from completion of brain irradiation.
* Females of childbearing potential as well as males and their partners must agree to use an effective form of contraception during the study and for 6 months following the last dose of study medication.

Exclusion Criteria:

* Clinically significant unrelated illness which would, in the judgment of the treating physician, compromise the patient's ability to tolerate the investigational agent or be likely to interfere with the study procedures or results.
* Patients with baseline corrected QT interval(QTc) > 480 msec.
* Known hypersensitivity to any of the components of irinotecan liposomes or prior hypersensitivity reactions to that class of drugs.
* Concomitant use of any other investigational or anticancer agent(s).
* Pregnant patients or patients who are breast feeding. Subjects capable of pregnancy (post menarche and not post-menopausal, defined as over 12 months since final menstrual period) must have a negative pregnancy test within 7 days prior to first dose.
* Other clinically significant malignant disease diagnosed within the previous 5 years, excluding intra-epithelial cervical neoplasia or non-melanoma skin cancer.
* Known persistent (> 4 weeks) ≥ Grade 2 neutropenia, ≥ Grade 2 thrombocytopenia or > Grade 3 anemia from prior cancer therapy.
* Other kinds of malignant tumors at the same time.

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 6 weeks
  To evaluate the maximum tolerated dose of weekly irinotecan liposomes for patients with relapsed or refractory Ewing sarcoma.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  To assess the preliminary response rate of irinotecan liposomes in patients with relapsed or refractory Ewing sarcoma.
Progression Free Survival (PFS) | 24 months
  To assess the preliminary progression free survival of irinotecan liposomes in patients with relapsed or refractory Ewing sarcoma.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shandong Cancer Hospital and Institute, Jina, Shandong
  - Peking University People's Hospital, Beijin
  - Peking University Shougang Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No